CLINICAL TRIAL: NCT03088501
Title: Participant Engagement and Retention Trial in a Public Hospital (PERTH): An RCT Protocol
Acronym: PERTH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PERTH RCT was nested within the MAASTHI birth cohort. PERTH study was stopped as MAASTHI has completed it's recruitment.
Sponsor: Public Health Foundation of India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LN0182
Record Dates: First submitted 2016-12-14; First posted 2017-03-23 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Intervention Study
Keywords: Birth cohort, follow-up, IVRS

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into each arm on a 1:1:1, using a computer-generated randomization list. Written allocation of assignments will be sealed in individual, sequentially numbered, non-resealable, opaque envelopes that will be used to allocate to the targeted number of participants.Once the participant is assigned to the arm, their unique respondent Identification Number ID(RID) and the arm to which they are allocated are recorded by the research assistants
Who Masked: Outcomes Assessor
Masking Description: After meeting inclusion criteria, consenting to participate and completing a baseline questionnaire, participants will be immediately assigned to the randomized study arm by the RA who will open one of the sequentially numbered envelopes to determine allocation. Before opening the envelope, the Respondent ID number will be written on the envelope. The assignment schedule will be kept in a locked filing cabinet in the study coordinator's office at the Indian Institute of Public Health. Research staff and pregnant women cannot be blinded because the intervention requires their participation; however, the data analyst will be blinded to the study arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interactive Voice Response System (Experimental): Through IVRS, women will receive a 2-3 minute call that informs them about their lab test, next follow-up visit, breastfeeding, introduction of solid foods, immunization, motor development, and sleep.
  Interventions: Behavioral: Interactive voice response system
- Mother and Baby Affairs (MBA) workshops (Experimental): This will involve antenatal workshop and counselling for parents.
  * Brief talk by health professionals.
  * Role-plays
  Interventions: Behavioral: Mother and baby affairs workshop
- Control Arm (No Intervention): The participants in this group do not get any specific interventions but would receive standard instructions to attend follow-up.

INTERVENTIONS:
Behavioral: Interactive voice response system — IVR allows the pregnant women, their family members to interact with a computer system using a telephone.Through IVR, women receive a 2-3 minute call that reminds them of lab test, their next follow-up visit and also provides information on child care attendance, breastfeeding, introduction of solid foods, motor development, and sleep.
  Arms: Interactive Voice Response System
Behavioral: Mother and baby affairs workshop — Mother and baby affairs workshop will involve antenatal workshop and counseling for parents. The intervention will involve brief talk by health professionals, quiz activities, role-plays on personal hygiene, nutritional food, institutional delivery, precautions at the time of delivery, caring for the baby, feeding of colostrum, homemade baby food, immunization, and family planning measures.
  Arms: Mother and Baby Affairs (MBA) workshops

SUMMARY:
MAASTHI (Maternal Antecedents of Adiposity Studying the Transgenerational role of Hyperglycaemia and Insulin) is a prospective birth cohort with the aim of assessing the effects of glucose levels in pregnancy on the risk of adverse infant outcomes, especially in predicting the possible risk markers of later chronic diseases. The recruitment of the pregnant women in MAASTHI has begun in the month of April 2016. Of the eligible pregnant women only 77% completed the oral glucose tolerance tests.The follow ups of mother and child are conducted at birth and annually during the year 1, 2, 3 and 4 of the child. Despite stringent adherence of including only the residents of the source population, nearly 13% of the women were lost to follow-ups at birth. In order to prevent further loss to follow-ups in subsequent visits, the investigators aim to explore whether interventions involving innovative Interactive Voice Response System (IVRS) and conducting mother and baby workshops can improve in the number pf women undergoing lab tests and subsequent follow-ups.

DETAILED DESCRIPTION:
Longitudinal cohort studies are important for the understanding of etiological mechanisms of underlying hypotheses. However, it is particularly challenging to sustain participation of subjects in follow up visits in birth cohorts, as the observation period spans over several years, making it vulnerable to lose tracking subjects for several reasons. These include change in location of residence and lack of interest in the later stages of the study. In India, the traditional practice of pregnant women leaving the study area to return to their maternal residence for delivery. Few groups belonging to ethnic minorities, with low family income or low education can be at higher risk of selective attrition. In the absence of high follow-up rate, the results from prospective cohort studies are can be biased. Such a bias can occur if the reason for the loss is related to the outcome under investigation. The cohort studies done in India have variable rates of loss to follow-up varying from, 14-82%. The barriers for retaining greater proportion of study participants can be due to several reasons. While a number of reviews have reported different ways of improving study participation, little is known about the effectiveness of specific retention strategies deployed in retention of mothers and infants in a birth cohort.

The proportion of pregnant women turning up for regular antenatal health checkups is poor in India. This is due to several reasons including lack of awareness, lack of social support, long waiting time, financial constraints and fear of hospital care. Evidence suggests that maternal education, husband's education, marital status, availability, cost, household income, women's employment, media exposure and previous obstetric history affects uptake of antenatal care services. According to National Family Health Survey (NFHS) (2014-15), only 55.5% of women in urban Bangalore had completed the required four antenatal care visits during pregnancy.

MAASTHI (Maternal Antecedents of Adiposity Studying the Transgenerational role of Hyperglycaemia and Insulin) is a prospective birth cohort with the aim of assessing the effects of glucose levels in pregnancy on the risk of adverse infant outcomes, especially in predicting the possible risk markers of later chronic diseases. The recruitment of the pregnant women in MAASTHI has begun in the month of April 2016. Of the eligible pregnant women only 77% completed the oral glucose tolerance tests despite offering the test free of cost and repeated reminders by the research team to get tested for gestational diabetes. After completion of OGTT, the follow ups of mother and child are conducted at birth and annually during the year 1, 2, 3 and 4 of the child. Despite stringent adherence of including only the residents of the source population, nearly 13% of the women were lost to follow-ups at birth. These women delivered in a different hospital mostly due to obstetric complications. Currently around 80 participants are recruited per month, with completion of all their records, anthropometry measurements, and Oral Glucose Tolerance Test (OGTT). Once the OGTT is done between 24-32 weeks of gestation, there is no further opportunity to meet them again till the delivery. The duration without contact increases the likelihood for attrition of future follow-ups. In the intervening period of initial contact and follow-up's, it is important that the research staff constantly engage with the participants through innovative methods. In order to improve the number of women undergoing OGTT and follow-ups, an intervention trial will be carried out that examines the role of innovative 1) IVR and 2)Mother and baby workshops during the intervening time period between baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women between 14 to 28 weeks of gestational age and those who plan to deliver in the study hospital and reside in the study location for the next five years. She must be able to speak Kannada, Hindi or English and should be willing to provide informed consent voluntarily. The participant must own or have sufficient access to a cell phone and should be able to operate a cell phone with a partner, relative, etc who stay with her.

Exclusion Criteria:

* Diabetes or Hepatitis B infection;
* HIV positivity;
* Pregnant women of other gestational ages

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the proportion of participants visiting the hospital for OGTT before 32 weeks of gestation. | 10 week
  Successful follow-up assessment will be defined as completion of lab tests of mother within the designated time of 32 weeks of gestation. Response rate will be estimated as the number of women who complete lab tests done by research staff divided by the total number of women who completed 32 weeks of gestation. Loss to follow up rate will be measured as the number of women who missed lab tests divided by the total number of women who completed 32 weeks of gestation during the corresponding study time period in the study population. Time frame is calculated based on the start of the intervention at 22 week of gestation to the time when the mother's gestational age is 32 weeks, which is a total duration of 10 weeks.
The proportion of participants who successfully complete follow-up assessment within one week of delivery | 18 week
  Those who successfully complete, follow-up assessment within one week of delivery. Successful follow-up assessment will be defined as completion of follow-up questionnaire and anthropometry within the designated time of one week from the date of delivery. Follow-up rate will be estimated as the numbers of follow ups done by research staff divided by the total number of eligible live births due in the corresponding time period in the study population. The loss to follow up rate will be measured as the number of missed follow-ups divided by the total number of eligible live births due in the corresponding time period in the study population. The time frame is calculated based on the start of the intervention at 22 weeks of gestation to 40 weeks at the time of delivery, which is the duration of 18 weeks.
The proportion of participants who successfully complete second follow-up assessment when the infant is 3.5 month old. | 32 week
  Successful follow-up assessment will be defined as completion of follow-up questionnaire and anthropometry of mother and child within the designated time of 3.5 months ±15 days since the date of birth. Follow-up rate will be estimated as the number of 3.5 months follows ups done by research staff divided by the total number of 3.5-month-old infants during the corresponding study time period in the study population. The loss to follow up rate will be measured as the number of missed follow-ups divided by the total number of 3.5-months-old infants during the corresponding study time period in the study population. The time frame is calculated based on the start of the intervention at 22 weeks of gestation to the time when the infant is 3.5 months old(14 weeks) which is a total duration of 32 weeks.

SECONDARY OUTCOMES:
The secondary outcome involves cost-benefit analysis of the IVRS and MBA workshop | 40 week
  An economic evaluation of the intervention package in improving successive health visits compared to a control group will be done. A cost-effectiveness analysis will be done by assessing the balance between costs of the intervention and effects of improved visits from a healthcare provision perspective. Costs for all separate actions and time used by all individual healthcare professionals will be mapped including the costs towards the workshop program, costs for the IVRS and all other materials. The costs involved in the intervention package and the benefits achieved will be compared with those of control arm.Time frame: cost effective analysis will be done within 8 weeks after the 3.5 month follow-up.(32 week+8 week=40 week)

CONTACTS AND LOCATIONS:
Locations (1):
- Sri rampura Referral Hospital, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
There is no drug or device being tested. This trial involves testing out the behavioural intervention in comparison with phone based technology for interactive voice based response to increase the follow-up of pregnant women.

REFERENCES:
- [Derived] Babu GR, Karthik M, Ravi D, Ana Y, Shriyan P, Hasige KK, Deshpande K, Siddlingaiah LB, Kinra S, Murthy GVS. What makes the pregnant women revisit public hospitals for research? Participant engagement and retention trial in a public hospital (PERTH): an RCT protocol. BMC Pregnancy Childbirth. 2018 Sep 12;18(1):369. doi: 10.1186/s12884-018-2000-1. PMID 30208868
- Available data/document: Protocol of the birth cohort: PMID: PMC5065083 — https://bmcpregnancychildbirth.biomedcentral.com/articles/10.1186/s12884-016-1088-4 — The proposed randomized controlled trial is nested within the MAASTHI Birth cohort in order to improve the follow-up rates.